CLINICAL TRIAL: NCT01943942
Title: Open, Two Periods, Two Treatments, Two Sequences, Cross-over, Randomized Study With Single Dosage of Two Oral Preparations Containing Montelukast 10 mg (Product of GlaxoSmithKline México, S.A. de C.V. vs. Singulair, Merck Sharp & Dohme de México, S.A. de C.V.)in Fasting Healthy Volunteers
Brief Title: Bioequivalence Study of Montelukast 10 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117015
Record Dates: First submitted 2012-11-28; First posted 2013-09-17 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Mexico; Montelukast; Pharmacokinetics; Bioequivalence
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (reference)/ B (test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Montelukast 10 mg
- B (test)/ A (reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Montelukast 10 mg

INTERVENTIONS:
Drug: Montelukast 10 mg — Reference product
  Other Names: Singulair; Merck Sharp & Dohme
Drug: Montelukast 10 mg — Test product

SUMMARY:
The objective of this study was to confirm if two formulations of montelukast tablets are bioequivalent.

Test product was Montelukast (10 mg tablets; GlaxoSmithKline) and reference product Singulair (10 mg tablets; Merck Sharp & Dohme). The single dosage was one tablet.

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fasting conditions.

The population was composed of 32 healthy volunteers, both genders, adults between 18-50 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

Free will participation according to Mexican regulation, Helsinki Declaration, and Good Clinical Practice.

Healthy, between 18 and 50 years. Body Mass Index between 19 and 27 In good health by complete medical history and laboratory tests. Blood pressure 130-90/ 90-60 mm Hg; heart rate 55-100 beat per minute, respiratory rate 14-20 movements per minute.

Laboratory tests +/- 10% of normal interval (blood cytology, blood chemistry 27 elements, Hepatitis B and C antigens, HIV, urinalysis, anti-doping, pregnancy, electrocardiogram) -

Exclusion Criteria:

Alteration of vital signs Not complying with inclusion criteria History of cardiovascular, kidney, hepatic, muscular, metabolic, gastrointestinal (including constipation), neurologic, endocrine, hematopoietic (any kind of anemia), asthma, mental or organic disease. Those suffering from muscular trauma 21 days before the beginning of the study.

Requirement of any kind of medication during the course of the study, except study medication.

History of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer. Exposure to medications known as inducers or inhibitors of hepatic enzymes or administration of potentially toxic medication in the 30 days before the study beginning.

Administration of any medication in the 14 days or 5 half-lives (whatever longer) previous to the beginning of the study.

Hospitalization for any cause in the seven months before the beginning of the study.

Administration of investigational drugs in the 60 days before the study. Allergy to any antibiotics or non-steroidal anti-inflammatory analgesics. Alcohol ingestion or intake of beverages containing xanthines (coffee, tea, cocoa, chocolate, mate, cola drinks) or ingestion of charcoal grilled food or grapefruit or orange juice in the 72 hours before the hospitalization or tobacco smoking in the 72 hours before the beginning of the study.

Blood donation or loss => 450 ml in the 60 days before the beginning of the study.

History of drug or alcohol abuse. Special diet requirement, for instance vegetarian diet. Inability to understand nature, aims, and possible consequences of the study. Non-cooperative attitude during the study. Positive anti-doping or pregnancy test. Breast-feeding. Females on contraceptive hormonal treatment.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05-16 (Actual); Primary Completion 2010-05-26 (Actual); Study Completion 2010-05-26 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of montelukast | 0.0, 0.5, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 4.5, 5, 6, 8, 10, 12, 15, and 18 hours postdosage
  Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of montelukast | 0.0, 0.5, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 4.5, 5, 6, 8, 10, 12, 15, and 18 hours postdosage
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 117015 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117015?search=study&study_ids=117015#rs